CLINICAL TRIAL: NCT00832962
Title: Effectiveness of Routine Fetal RhD Genotyping for RhD- Pregnant Women
Brief Title: Routine Fetal RhD Genotyping for RhD- Pregnant Women
Acronym: GENIFERH
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P 060410; IC 0606
Record Dates: First submitted 2009-01-13; First posted 2009-01-30 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Rhesus Negative Pregnant Women
Keywords: Rhesus D; Anti-D allo-immunization; Fetal RHD genotyping; anti-D immunoglobulins; anti-D prophylaxis
MeSH Terms: interventions — Genotype

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood sample (0.5 ml)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Adult Rh negative pregnant patients from 7 selected centers (SAINT ANTOINE hospital, CHU Marseille, CHU Nantes, CHU Lille, LOUIS MOURIER Hospital, SAINT VINCENT-PAUL Hospital, CH POISSY)
  Interventions: Genetic: Genotyping
- 2: Adult Rh negative pregnant patients from 6 selected centers (Tenon hospital, Jean VERDIER Hospital, La Pitie-Salpetriere Hospital, Cochin Hospital, Robert Debre Hospital, BICHAT Hospital)
  Interventions: Other: Usual prophylaxis

INTERVENTIONS:
Genetic: Genotyping — Whole blood sample
  Groups: 1
Other: Usual prophylaxis — Prophylactic anti-RhD
  Other Names: Prophylactic anti-RhD
  Groups: 2

SUMMARY:
The study is divided in two sub-studies. The first one is an economical and performance comparison between two antenatal management strategies of RhD negative pregnant women: the first one will comprise non invasive RhD fetal typing during the second trimester of pregnancy (GENIFERH 1 RhD typing group), and the second will be a conventional management, i.e. without RHD fetal typing (GENIFERH 1 control group). The two groups will consist of 13 maternity wards spread over French territory. The second study (GENIFERH 2) is an evaluation of RhD fetal typing diagnostic performance and biological feasibility in routine antenatal practice with development of knew technical support; it will be based on more than 3500 fetal genotypings performed during one year by the five laboratories participating at the two studies.

DETAILED DESCRIPTION:
Alloimmunisation against the RhD (RH) red cell surface antigen is the commonest cause of haemolytic disease of the fetus and newborn. It can be avoided by anti D immunoglobulin administration (RhIg). At the end of year 2005, new recommendations about anti-D prophylaxis in France proposed that all RhD negative pregnant women should be given anti-D immunoglobulin at 28 weeks' gestation. However, about one third of these women would be carrying an RhD negative fetus and would receive the treatment unnecessarily. A non-invasive fetal RHD typing kit, CE labelled since June 2007, is available and could be proposed to all RhD negative pregnant women. Applicable from the end of the first trimester of pregnancy on fetal DNA isolated from maternal plasma, this assay allows RhIg to be specifically injected to unsensitized pregnancies with RhD positive fetus only, and to promote the use of antenatal RhIg prophylaxis in a rational approach with economical and ethical impact.The study is divided in two sub-studies. The first one is an economical and performance comparison between two antenatal management strategies of RhD negative pregnant women: the first one will comprise non invasive RhD fetal typing during the second trimester of pregnancy (GENIFERH 1 RhD typing group), and the second will be a conventional management, i.e. without RHD fetal typing (GENIFERH 1 control group). The two groups will consist of 13 maternity wards spread over French territory. The second study (GENIFERH 2) is an evaluation of RhD fetal typing diagnostic performance and biological feasibility in routine antenatal practice with development of knew technical support; it will be based on more than 3500 fetal genotypings performed during one year by the five laboratories participating at the two studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult Rh negative pregnant patients ( ≥ 18 years)
* Valid and confirmed result of Rh D negative status.(one copy saved into the obstetrical records)
* Absence of actively produced anti-D antibody as shown on laboratory examination of a blood sample taken within the first trimester of pregnancy.
* Evolving pregnancy at the time of inclusion in the study ( between 8 and 26 gestation weeks as confirmed by early sonography).
* Absence of a previous invasive fetal RHD genotyping ( chorionic villous sampling, amniocentesis).
* Patient having signed an informed consent for the study.
* Inclusion and delivery expected in the same maternity ward
* Patient affiliated to a social security regimen.

Exclusion Criteria:

* Evolving pregnancy seen for the first time after 26 gestation weeks.
* Poor understanding of the objectives of the study ( language barrier, ...)
* Delivery expected in a maternity ward not participating at the study.
* Fetal RHD invasive genotyping performed during early pregnancy on amniotic fluid or chorionic villus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Rh negative pregnant women followed in the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 2532 (Actual)
Dates: Start 2009-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
cost-effectiveness of the two strategies of antenatal management by comparing the rate of RhD negative women eligible for receiving RHIG that would have not receive prophylactic anti-RhD in the two populations, the one with fetal RHD typing and the other | At the end of the study

SECONDARY OUTCOMES:
Assessment of the applicability of non invasive fetal RHD typing in the antenatal management of unimmunized Rh-negative pregnant patients in different settings. | At the end of the study
performance assessment of high throughput fetal RHD genotyping in hospital laboratories. | At the end of the study
Evaluation of the technical support needed to realize high throughput fetal RHD genotyping by authorized laboratories. | At the end of the study
Development and diffusion of external quality controls for non invasive fetal RHD genotyping. | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Yves BROSSARD, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Saint Antoine, Paris, France

REFERENCES:
- [Background] Branger B, Winer N. [Epidemiology of anti-D allo-immunization during pregnancy]. J Gynecol Obstet Biol Reprod (Paris). 2006 Feb;35(1 Suppl):1S87-1S92. French. PMID 16495833
- [Background] Parant O. [Comparison of the efficacy of different methods for the prevention of anti-D allo-immunization during pregnancy: targeted strategy limited to risk situations or associated with systematic prevention in the 3rd trimester]. J Gynecol Obstet Biol Reprod (Paris). 2006 Feb;35(1 Suppl):1S93-1S103. French. PMID 16495834
- [Background] Bennett PR, Le Van Kim C, Colin Y, Warwick RM, Cherif-Zahar B, Fisk NM, Cartron JP. Prenatal determination of fetal RhD type by DNA amplification. N Engl J Med. 1993 Aug 26;329(9):607-10. doi: 10.1056/NEJM199308263290903. PMID 8341334
- [Background] Aubin JT, Le Van Kim C, Mouro I, Colin Y, Bignozzi C, Brossard Y, Cartron JP. Specificity and sensitivity of RHD genotyping methods by PCR-based DNA amplification. Br J Haematol. 1997 Aug;98(2):356-64. doi: 10.1046/j.1365-2141.1997.2193040.x. PMID 9266934
- [Background] Lo YM, Corbetta N, Chamberlain PF, Rai V, Sargent IL, Redman CW, Wainscoat JS. Presence of fetal DNA in maternal plasma and serum. Lancet. 1997 Aug 16;350(9076):485-7. doi: 10.1016/S0140-6736(97)02174-0. PMID 9274585
- [Background] Lo YM, Tein MS, Lau TK, Haines CJ, Leung TN, Poon PM, Wainscoat JS, Johnson PJ, Chang AM, Hjelm NM. Quantitative analysis of fetal DNA in maternal plasma and serum: implications for noninvasive prenatal diagnosis. Am J Hum Genet. 1998 Apr;62(4):768-75. doi: 10.1086/301800. PMID 9529358
- [Background] Brossard Y, Sender A, Cartron JP, Huchet J, Pinon F, Blot P, David G. [Value of RHD fetal genotyping in the prevention of anti-D immunization]. Bull Acad Natl Med. 2001;185(2):329-36. French. PMID 11474588
- [Background] Faas BH, Beuling EA, Christiaens GC, von dem Borne AE, van der Schoot CE. Detection of fetal RHD-specific sequences in maternal plasma. Lancet. 1998 Oct 10;352(9135):1196. doi: 10.1016/s0140-6736(05)60534-x. No abstract available. PMID 9777844
- [Background] Rouillac-Le Sciellour C, Puillandre P, Gillot R, Baulard C, Metral S, Le Van Kim C, Cartron JP, Colin Y, Brossard Y. Large-scale pre-diagnosis study of fetal RHD genotyping by PCR on plasma DNA from RhD-negative pregnant women. Mol Diagn. 2004;8(1):23-31. doi: 10.1007/BF03260044. PMID 15230639
- [Background] Colin Y, Cherif-Zahar B, Le Van Kim C, Raynal V, Van Huffel V, Cartron JP. Genetic basis of the RhD-positive and RhD-negative blood group polymorphism as determined by Southern analysis. Blood. 1991 Nov 15;78(10):2747-52. PMID 1824267
- [Background] Singleton BK, Green CA, Avent ND, Martin PG, Smart E, Daka A, Narter-Olaga EG, Hawthorne LM, Daniels G. The presence of an RHD pseudogene containing a 37 base pair duplication and a nonsense mutation in africans with the Rh D-negative blood group phenotype. Blood. 2000 Jan 1;95(1):12-8. PMID 10607679
- [Background] Geifman-Holtzman O, Grotegut CA, Gaughan JP. Diagnostic accuracy of noninvasive fetal Rh genotyping from maternal blood--a meta-analysis. Am J Obstet Gynecol. 2006 Oct;195(4):1163-73. doi: 10.1016/j.ajog.2006.07.033. PMID 17000250
- [Background] Lo YM, Hjelm NM, Fidler C, Sargent IL, Murphy MF, Chamberlain PF, Poon PM, Redman CW, Wainscoat JS. Prenatal diagnosis of fetal RhD status by molecular analysis of maternal plasma. N Engl J Med. 1998 Dec 10;339(24):1734-8. doi: 10.1056/NEJM199812103392402. PMID 9845707
- [Background] Finning K, Martin P, Daniels G. A clinical service in the UK to predict fetal Rh (Rhesus) D blood group using free fetal DNA in maternal plasma. Ann N Y Acad Sci. 2004 Jun;1022:119-23. doi: 10.1196/annals.1318.019. PMID 15251949
- [Background] van der Schoot CE. Molecular diagnostics in immunohaematology. Vox Sang. 2004 Jul;87 Suppl 2:189-92. doi: 10.1111/j.1741-6892.2004.00481.x. No abstract available. PMID 15209914
- [Background] Cortey A, Brossard Y, Beliard R, Bourel D. [Prevention of fetomaternal rhesus-D allo-immunization. Perspectives]. J Gynecol Obstet Biol Reprod (Paris). 2006 Feb;35(1 Suppl):1S119-1S122. French. PMID 16495837
- [Background] Zimmermann B, El-Sheikhah A, Nicolaides K, Holzgreve W, Hahn S. Optimized real-time quantitative PCR measurement of male fetal DNA in maternal plasma. Clin Chem. 2005 Sep;51(9):1598-604. doi: 10.1373/clinchem.2005.051235. Epub 2005 Jul 14. PMID 16020496
- [Background] Chan KC, Ding C, Gerovassili A, Yeung SW, Chiu RW, Leung TN, Lau TK, Chim SS, Chung GT, Nicolaides KH, Lo YM. Hypermethylated RASSF1A in maternal plasma: A universal fetal DNA marker that improves the reliability of noninvasive prenatal diagnosis. Clin Chem. 2006 Dec;52(12):2211-8. doi: 10.1373/clinchem.2006.074997. Epub 2006 Oct 26. PMID 17068167
- [Background] Daniels G, van der Schoot CE, Olsson ML. Report of the Second International Workshop on molecular blood group genotyping. Vox Sang. 2007 Jul;93(1):83-8. doi: 10.1111/j.1423-0410.2007.00926.x. PMID 17547570
- [Background] Hayes RJ, Bennett S. Simple sample size calculation for cluster-randomized trials. Int J Epidemiol. 1999 Apr;28(2):319-26. doi: 10.1093/ije/28.2.319. PMID 10342698
- [Derived] Darlington M, Carbonne B, Mailloux A, Brossard Y, Levy-Mozziconacci A, Cortey A, Maoulida H, Simon T, Rousseau A, Durand-Zaleski I; GENIFERH1 Study Group. Effectiveness and costs of non-invasive foetal RHD genotyping in rhesus-D negative mothers: a French multicentric two-arm study of 850 women. BMC Pregnancy Childbirth. 2018 Dec 14;18(1):496. doi: 10.1186/s12884-018-2114-5. PMID 30547830